CLINICAL TRIAL: NCT04073225
Title: Optimizing Cognitive, Environmental, and Neuromotor Stimulation in Traumatic Brain Injury (OCEANS-TBI)
Brief Title: Optimizing Cognitive, Environmental, and Neuromotor Stimulation in Traumatic Brain Injury
Acronym: OCEANS-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00218229
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury; Dementia Alzheimers; Military Activity
Keywords: veteran
MeSH Terms: conditions — Brain Injuries, Traumatic; Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MindPod Dolphin Arm (Experimental): Bandit the Dolphin provides an oceanic environment in which the individual's arm movements control a simulated dolphin. The neuromotor effects of this game have been designed to be used in the clinical setting to rehabilitate arm and hand function following stroke.
  Interventions: Device: MindPod Dolphin
- 10 Keys to Healthy Aging (Active Comparator): The "10 Keys"™ to Healthy Aging Program is designed to teach older adults how to reduce the risk of disease over the aging process by promoting healthy lifestyle changes with the most recent established scientific guidelines.
  Interventions: Behavioral: 10 Keys to Healthy Aging

INTERVENTIONS:
Device: MindPod Dolphin — The immersive video game being tested in this study is called Bandit the Dolphin, developed by neurologist Dr. John Krakauer, and engineers in the Brain, Learning, Animation, and Movement Lab at Johns Hopkins. Bandit the Dolphin provides an oceanic environment in which the individual's arm movements control a simulated dolphin. The neuromotor effects of this game have been designed to be used in the clinical setting to rehabilitate arm and hand function following stroke. The game has further been modified to a Microsoft Kinect-based system and piloted for play in non-laboratory settings among community-dwelling adults. The game offers a unique combination of skilled arm movements plus varying levels of cognitive challenge. In this way, the individual's arms are challenged the same way the legs would be when walking in a complex, outdoor environment. Importantly, the participant "plays" while standing, thus engaging the whole body in this novel multi-sensorial experience.
  Other Names: Bandit the Dolphin
  Arms: MindPod Dolphin Arm
Behavioral: 10 Keys to Healthy Aging — The "10 Keys"™ to Healthy Aging Program in an evidence-based program that originated from the University of Pittsburgh Center for Aging and Population Health. This educates and empowers older adults to reach personal goals and help others to so in the community as well. It is designed to teach older adults how to reduce the risk of disease over the aging process by promoting healthy lifestyle changes with the most recent established scientific guidelines. The 10 Keys program also aims to empower individuals to be health ambassadors in the individual's own families and communities, teaching individuals to 'Share the Wealth on Health'. Participants will work towards personal health goal(s) adapted to the participant's lifestyle and abilities.
  Arms: 10 Keys to Healthy Aging

SUMMARY:
Patients with a history of traumatic brain injury (TBI) are at elevated risk for Alzheimer's disease and related dementias (ADRD). Improvements in TBI treatment may mitigate this risk. Complex motor activities, which combine physical and cognitive demands, have been shown to have well established neurocognitive benefits. This study seeks to address the need for novel TBI interventions optimized for adults with history of TBI by determining the effectiveness of an immersive computer game designed to integrating complex cognitive-motor interventions.

DETAILED DESCRIPTION:
Patients with a history of traumatic brain injury (TBI) are at elevated risk for Alzheimer's disease and related dementias (ADRD). Improvements in TBI treatment may mitigate this risk. The treatment of TBI, especially for those with chronic neuropsychiatric sequelae, is moving toward multi-modal approaches that include non-pharmacological interventions such as exercise and cognitive enrichment. Complex motor activities, which combine physical and cognitive demands, have been shown to have well established neurocognitive benefits. However, there are a lack of cognitive enhancing interventions that utilize these complex motor activities. Many adults with history of TBI face significant barriers to engaging in physical activity which limit the adults' ability to participate in many neurocognitive interventions. This study seeks to address the need for novel TBI interventions optimized for adults with history of TBI by determining the effectiveness of an immersive computer game designed to integrating complex cognitive-motor interventions. During this proposed 12-month study involving patients with history of TBI (n=66) the investigators will examine cognition, independent function, mood and ADRD related brain biomarkers after 12 weeks of a randomized intervention, as well as 9 months post-intervention to assess for durability of any benefits. The investigators hypothesize that complex motor activities will improve cognitive health in adults with a history of TBI and that promising results would have implications for early intervention for those at risk for Mild Cognitive Impairment and ADRD.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* 40 years of age and older
* History of at least one remote TBI (>3 years ago) of mild and moderate severity as diagnosed by Veteran's Affairs / Department of Defense (VA/DoD) criteria.
* Ability to perform most independent activities of daily living without physical assistance (e.g., no canes or walkers because person needs both hands to participate); Chedoke Arm and Hand Activity Inventory - mean score >5, indicating modified or complete independence in hand and arm functioning.
* Ability to dedicate 3 hours per week for about 12 weeks-approximately 20 to 26 hours of total time-to the intervention study.
* Ability to give informed consent and understand the tasks involved

Exclusion Criteria:

* Presence of cognitive impairment based on a Mini-Mental State Exam (MMSE) score ≤ 24.
* Presence of diseases associated with gross motor abnormalities that restrict ambulation (e.g., stroke with paresis, multiple sclerosis, amyotrophic lateral sclerosis, cerebellar or spinal cord disorders, peripheral nerve disorders, severe rheumatic or osteoarthritic disorders, limb amputation)
* Untreated major mental illness that may preclude successful completion of the study (e.g., major depressive disorder, anxiety disorders, etc.)
* History of physical or neurological condition that interferes with study procedures or assessment of motor function (e.g., epilepsy, severe arthritis, severe neuropathy, Parkinson's disease).
* Current diagnosis of color blindness.
* Social or personal circumstances that interfere with ability to complete 12-14 weeks of training sessions and follow-up evaluation.
* Inability to sit in a chair or stand and perform upper limb exercises for one hour at a time.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew E Peters, MD, Principal Investigator — Johns Hopkins University; Michelle C Carlson, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment sources included Johns Hopkins Alzheimer's Disease Research Center (ADRC), Bayview Community Psychiatry Program (CPP), Johns Hopkins Community Physicians (JHCP), JHCP Clinic Champion: advertises study in JHCP, Clinical Connection, ClinicalTrials.gov, ResearchMatch.org, MyChart, and newsletters/flyers.
Period: Overall Study
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging
Started | 14 | 9
Completed | 10 | 6
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (8.9) | 57.6 (13.3) | 59.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 9 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Executive Functioning as Assessed by the Trail Making Test
Description: The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two timed parts (Part A and B) in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. Our primary measure was the difference in time (seconds) taking to complete Part B subtracted by Part A, which is an indicator of task-switching.
Time Frame: Baseline, 12 weeks
Population: One participant was excluded due to missing data at both baseline and 12 week visits.
Measure: Mean (95% Confidence Interval); unit: change in seconds
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging
Number analyzed (Participants) | 13 | 9
change in seconds | -9.2 [-51.5 to 33.1] | 24.7 [-27.4 to 76.7]
Statistical Analysis 1: Comparison: MindPod Dolphin Arm vs 10 Keys to Healthy Aging; Mixed effects models were fit including fixed effects for intervention arm, visit (baseline, 12 week) and intervention by visit interaction; and random intercepts and slopes for each participant; Test type: Superiority; p = .323, Mixed Models Analysis; Mean Difference (Net) = -33.8, 95% CI 2-sided [-100.9 to 33.2]

2. Primary Outcome: Change in Executive Functioning as Assessed by the Stroop Test
Description: The Stroop Test is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. Our primary measure was the Stroop Effect (i.e., reaction time (milliseconds) for incongruent trials subtracted by reaction time for congruent trials).
Time Frame: Baseline, 12 weeks
Population: One participant was excluded due to missing data at both baseline and 12 week visits.
Measure: Mean (95% Confidence Interval); unit: change in milliseconds
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging
Number analyzed (Participants) | 13 | 9
change in milliseconds | -49.5 [-103.3 to 4.2] | 31.8 [-32.6 to 96.2]
Statistical Analysis 1: Comparison: MindPod Dolphin Arm vs 10 Keys to Healthy Aging; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .057, Mixed Models Analysis; Mean Difference (Net) = -81.3, 95% CI 2-sided [-165.2 to 2.5]

3. Primary Outcome: Change in Processing Speed Score as Assessed by the Pattern Comparison Test
Description: This test measures speed of processing by asking participants to discern whether two side-by-side pictures are the same or not. The processing speed score was the total number of trials completed correctly within the specified time limit.
Time Frame: Baseline, 12 weeks
Population: One participant was excluded due to missing data at both baseline and 12 week visits.
Measure: Mean (95% Confidence Interval); unit: trials
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging
Number analyzed (Participants) | 13 | 9
trials | 2.0 [0.1 to 4.0] | -1.0 [-3.4 to 1.3]
Statistical Analysis 1: Comparison: MindPod Dolphin Arm vs 10 Keys to Healthy Aging; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .047, Mixed Models Analysis; Mean Difference (Net) = 3.1, 95% CI 2-sided [0.03 to 6.08]

4. Primary Outcome: Change in Verbal Learning as Assessed by the Rey Auditory Verbal Learning Test (RAVLT)
Description: The investigators will assess for change in verbal learning using the RAVLT. The RAVLT is a neuropsychological assessment designed to evaluate verbal memory in patients, 16 years of age and older. The RAVLT can be used to evaluate the nature and severity of memory dysfunction and to track changes in memory function over time. The test is designed as a list-learning paradigm in which the patient hears a list of 15 nouns and is asked to recall as many words from the list as possible. Our primary measure was the number of words correctly recalled after a long delay (20 minutes), an indicator of long-term verbal memory.
Time Frame: Baseline, 12 weeks
Population: One participant was excluded due to missing data at both baseline and 12 week visits.
Measure: Mean (95% Confidence Interval); unit: words
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging
Number analyzed (Participants) | 13 | 9
words | 1.5 [0.2 to 2.7] | 0.9 [-0.6 to 2.4]
Statistical Analysis 1: Comparison: MindPod Dolphin Arm vs 10 Keys to Healthy Aging; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .565, Mixed Models Analysis; Mean Difference (Net) = .59, 95% CI 2-sided [-1.4 to 2.6]

5. Primary Outcome: Change in Physical Mobility Outcome as Assessed by the Short Physical Performance Battery
Description: The Short Physical Performance Battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. We measured the change in SPPB score from baseline to 12-week post-intervention follow-up assessments. Total score of 0 to 12, with a higher score indicating better physical function.
Time Frame: Baseline, 12 weeks
Population: There were 10 intervention participants and 6 control group participants that had data collected at both baseline and post-intervention 12-week follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging
Number analyzed (Participants) | 10 | 6
score on a scale | 0.67 (1.03) | -0.60 (1.83)
Statistical Analysis 1: Comparison: MindPod Dolphin Arm vs 10 Keys to Healthy Aging; Test type: Superiority; p = 0.147, t-test, 2 sided; Mean Difference (Net) = 1.27, 95% CI 2-sided [-0.50 to 3.03], Standard Error of Mean 0.825

6. Primary Outcome: Change in Brain Magnetic Resonance Imaging (MRI) Hippocampal Volume (mm3)
Description: Brain volumetrics will be calculated using a Philips 3 Tesla (T) head-only scanner using established methods. Hippocampal volumes were automatically segmented using Freesurfer and was summed across both hemispheres to calculate total volume. Change in total hippocampal volume from baseline to 12 weeks was used as the primary measure.
Time Frame: Baseline, 12 weeks
Population: Nine participants who had both baseline and 12 week MRI data were included in this analysis.
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging
Number analyzed (Participants) | 5 | 4
mm^3 | -109.7 (63.1) | -10.3 (192.2)
Statistical Analysis 1: Comparison: MindPod Dolphin Arm vs 10 Keys to Healthy Aging; We conducted t-tests of differences in volumetric change comparing intervention to control arms; Test type: Superiority; p = .605, t-test, 2 sided; Mean Difference (Net) = 99.4, 95% CI 2-sided [-334.3 to 533.0]

7. Primary Outcome: Change in Brain Magnetic Resonance Imaging (MRI) Amygdala Volume (mm3)
Description: Brain volumetrics will be calculated using a Philips 3 Tesla (T) head-only scanner using established methods. Amygdala volumes were automatically segmented using Freesurfer and were summed across both hemispheres to calculate total volume. Change in total amygdala volume from baseline to 12 weeks was used as the primary measure.
Time Frame: Baseline, 12 weeks
Population: Nine participants who had both baseline and 12 week MRI data were included in this analysis.
Measure: Mean (Standard Error); unit: mm3
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging
Number analyzed (Participants) | 5 | 4
mm3 | 67.1 (181.1) | -63.7 (148.8)
Statistical Analysis 1: Comparison: MindPod Dolphin Arm vs 10 Keys to Healthy Aging; We conducted t-tests of differences in volumetric change comparing intervention to control arms; Test type: Superiority; p = .590, t-test, 2 sided; Mean Difference (Net) = 130.8, 95% CI 2-sided [-259.7 to 248.6]

8. Secondary Outcome: Change in Time (Minutes) Spent Outside Home as Assessed by the Apple Watch GPS
Description: The investigators will assess time spent outside the home from an Apple Watch GPS. Time spent out of home is measured by summing total duration spent in latitude/longitude coordinates that fall outside of a 120 meter radial buffer around the participant's home address.
Time Frame: Baseline, 12 weeks
Population: There were 10 intervention group participants and 6 control group participants that had data collected for time spent outside of home at both baseline and 12-week post-intervention assessments.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging
Number analyzed (Participants) | 10 | 6
minutes | 59.99 (172.65) | 35.27 (60.09)
Statistical Analysis 1: Comparison: MindPod Dolphin Arm vs 10 Keys to Healthy Aging; Test type: Superiority; p = .743, t-test, 2 sided; Mean Difference (Net) = -24.72, 95% CI 2-sided [-183.11 to 133.68], Standard Error of Mean 73.85

9. Secondary Outcome: Change in Depressive Symptoms as Assessed by the Patient Health Questionnaire - 9 (PHQ-9)
Description: The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. The PHQ-9 incorporates Diagnostic and Statistical Manual-IV depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool. Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe (total score range of 0-27). Higher score worse/more severe symptoms.
Time Frame: Baseline, 12 weeks
Population: There were 10 intervention and 4 control group participants with available data for PHQ-9 at both baseline and 12-week post-intervention assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging
Number analyzed (Participants) | 10 | 4
score on a scale | 0.10 (4.72) | -1 (6.68)
Statistical Analysis 1: Comparison: MindPod Dolphin Arm vs 10 Keys to Healthy Aging; Test type: Superiority; p = 0.731, t-test, 2 sided; Mean Difference (Net) = -1.1, 95% CI 2-sided [-7.91 to 5.71], Standard Error of Mean 3.13

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, approximately 12 months
Arm/Group | MindPod Dolphin Arm | 10 Keys to Healthy Aging
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/9
Other Adverse Events (participants affected / at risk) | 0/14 | 0/9

LIMITATIONS AND CAVEATS:
A significant limitation of the study was the small sample size. This limited enrollment fell short of the target number needed to achieve sufficient statistical power, which reduced the reliability of the results and limited the ability to detect meaningful intervention effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT04073225/Prot_SAP_000.pdf